CLINICAL TRIAL: NCT03979768
Title: Risk Assessment and HaemoglobinA1c (HbA1c) -Measurement in Community Pharmacies to Identify People With Undiagnosed Type 2 Diabetes
Brief Title: Risk Assessment of Type 2 Diabetes in Pharmacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016/808
Record Dates: First submitted 2019-03-22; First posted 2019-06-07 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: Eight community pharmacies offered a diabetes risk assessment including a diabetes risk assessment test only, while 11 community pharmacies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risk Assessment Only pharmacies (RTO-group) (Experimental): Offered a diabetes risk assessment service without any blood sample testing.
  Interventions: Other: Diabetes risk assessment service in Norwegian community pharmacies
- HbA1c-group /pharmacies (Experimental): Offered a diabetes risk assessment service including a measurement of Haemoglobin A1c (HbA1c) to the people with a high risk of developing type 2 diabetes on the risk assessment form (The Finnish Diabetes Risc Score (FINDRISC) to those with a western background, and Leicester Risk Assessment (LRA) form for those with a non-western background.
  Interventions: Other: Diabetes risk assessment service in Norwegian community pharmacies

INTERVENTIONS:
Other: Diabetes risk assessment service in Norwegian community pharmacies — Two pharmacists at each pharmacy were trained to perform risk assessments and counselling. During six months, pharmacy customers equal or above 45 years old, wishing to participate contacted the pharmacy staff. Participants completed a validated diabetes risk test and a background questionnaire including a validated instrument for self-rated health.

SUMMARY:
Background: Due to lack of clear symptoms, type 2 diabetes can remain undetected for many years. Our aim was to explore the capacity of Norwegian community pharmacies to identify people at high risk of developing type 2 diabetes and the impact of the risk assessment service on self-rated health.

Methods: Nineteen community pharmacies were randomly allocated to a diabetes risk test only- group or Haemoglobin A1c (HbA1c) -group were the participants with a high risk of developing type 2 diabetes also received a HbA1c-measurement. Two pharmacists at each pharmacy were trained to perform risk assessments and counselling. The pharmacists at the 11 HbA1c pharmacies were also trained in how to perform the HbA1c- measurement. During six months, pharmacy customers equal or over 45 years old, wishing to participate contacted the pharmacy staff. Participants completed a validated diabetes risk test and a background questionnaire including a validated instrument for self-rated health. In the risk test only-group, participants with a high risk of developing type 2 diabetes were referred to their general practitioner for follow-up, while in the HbA1c-group, participants with HbA1c ≥ 48 mmol/ mol (6.5%) were referred to their general practitioner.

DETAILED DESCRIPTION:
Background: Due to lack of clear symptoms, type 2 diabetes can remain undetected for many years. Our aim was to explore the capacity of Norwegian community pharmacies to identify people at high risk of developing type 2 diabetes and the impact of the risk assessment service on self-rated health.

Methods: Nineteen community pharmacies were randomly allocated to a diabetes risk test only- group or Haemoglobin A1c (HbA1c) -group were the participants with a high risk of developing type 2 diabetes also received a HbA1c-measurement. Two pharmacists at each pharmacy were trained to perform risk assessments and counselling. The pharmacists at the 11 HbA1c pharmacies were also trained in how to perform the HbA1c- measurement. During six months, pharmacy customers equal or above 45 years old, wishing to participate contacted the pharmacy staff. Participants completed a validated diabetes risk test and a background questionnaire including a validated instrument for self-rated health. In the risk test only-group, participants with a high risk of developing type 2 diabetes were referred to their general practitioner for follow-up, while in the HbA1c-group, participants with HbA1c ≥ 48 mmol/ mol (6.5%) were referred to their general practitioner.

ELIGIBILITY:
Inclusion Criteria:

- age equal to or above 45 years old (increased from 18 years in the feasibility study), and being able to read and write Norwegian/English.

Exclusion Criteria:

- known diabetes, pregnancy and blood diseases that may affect measurement of Haemoglobin A1c (HbA1c).

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with undiagnosed type 2 diabetes | 2 months
  Number of Participants with undiagnosed type 2 diabetes

SECONDARY OUTCOMES:
Explore if there was any difference in the number of participants with a high risk of developing type 2 diabetes in the risk test only (RTO)- group and the group that also offered a HbA1c-measurement (HbA1c-group) | Baseline
  Find the number of participants with a high risk of developing type 2 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Aslaug Johanne Risøy, PhDCandidate, Principal Investigator — University of Bergen

IPD SHARING:
Plan to Share IPD: No